CLINICAL TRIAL: NCT01617499
Title: Physical Activity for Campus Employees
Acronym: PACE
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201109022
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Cardiovascular Disease
Keywords: physical activity; pedometer; worksite; wellness; cardiovascular; lifestyle program
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- University employees: Participants will include employees of Washington University in St. Louis. Recruitment will be directed to staff employees of the Central Fiscal Unit (CFU) on the Danforth campus.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — The worksite wellness program included cardiovascular health assessments, personal health reports, 8 weeks of pedometer-based walking and tracking activities, and weekly wellness sessions.

SUMMARY:
The aim of this pilot study is to evaluate the effects of a worksite wellness program on physical activity and cardiovascular disease risk factors among university employees. The investigators hypothesize that the proposed worksite wellness program will be effective for increasing daily physical activity and improving one or more cardiovascular disease risk factors among university employees.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) persists as the leading cause of mortality in the United States and accounts for 17 percent of the nation's overall health expenditures. Although the mortality rate of CVD has declined in recent years, the burden of disease remains high. Currently, 1 in 3 Americans has some form of CVD. Additionally, according to a recent policy statement published by the American Heart Association (AHA), 40% of the population is projected to have some form of CVD by 2030. Furthermore, the AHA has projected that the cost to treat CVD will triple by 2030. The prevalence and rising financial burden of CVD demonstrate the urgency for effective implementation of disease prevention strategies.

Evidence suggesting the majority of CVD is preventable through modifiable risk factor management continues to grow. Nonetheless, difficulty controlling modifiable risk factors remains an issue for many Americans. The magnitude of this challenge is supported by a study revealing that 78% of adults are candidates for at least one CVD prevention activity. Although national organizations have published a variety of disease prevention recommendations, widespread implementation of and adherence to preventative programs remain problematic. Consequently, a large proportion of the population is not receiving or participating in prevention strategies from which they may benefit. The full potential of reducing the nation's CVD burden cannot be achieved unless interventions are implemented on a larger scale, with reduced costs, and with increased initial and continued participation.

With approximately 130 million Americans currently employed, workplaces provide ideal environments for implementation of sizable, cost-effective CVD prevention programs. However, successful wellness programming remains a laborious, resource intensive challenge for employers. In 2004, a National Worksite Health Promotion Survey disclosed that less than 7% of U.S. employers offered worksite wellness programs. Furthermore, an estimated 25-30% of companies' annual medical costs are spent on employees with CVD risk factors.

In the proposed study, a worksite wellness program that includes health assessments, personal health reports, and pedometer-based tracking of physical activity will be offered to university employees. Participants will not be randomized to an intervention or control group. Rather, program components will be available to all enrolled participants, and each individual may choose whether to wear a pedometer, track their step counts, attend wellness sessions, and/or complete the health assessments. There is no prescribed intervention. Wellness sessions include educational information on lifestyle behaviors to promote cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* employee of Washington University in St. Louis

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of employees of Washington University in St. Louis. A convenience sample of staff employees located on the Danforth campus will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Daily Step Count (determined by pedometer) | Baseline, week 4, and week 8
  Daily step counts, as recorded by pedometers, will be self-reported by participants for 7 continuous days at 3 study time points: baseline, week 4, and week 8.

SECONDARY OUTCOMES:
Body weight | Baseline and week 9
  Body weight will be measured on a digital scale in the morning after an overnight fast. Shoes, jewelry, sweaters, jackets, belts, and hats will be removed and pockets will be emptied before the measurement is made.
Body Mass Index (BMI) | Baseline and week 9
  BMI will be computed as weight in kilograms divided by height in meters squared. Weight Status will be determined using standard CDC BMI categories.
Body Composition | Baseline and week 9
  Fat mass (kg), fat free mass (kg), and percentage body fat will be determined by bioelectrical impedance analysis using the InBody 520 analyzer.
waist circumference | Baseline and week 9
  Waist circumference will be measured at the border of the iliac crest using a Gulick II tape measure.
Blood Pressure | Baseline and week 9
  Systolic and diastolic blood pressure will be measured in duplicate in the right arm after 10 minutes of seated rest using the Omron HEM-907XL Professional Digital Blood Pressure Monitors (Omron Healthcare, Kyoto, Japan). One minute rest will be provided between the 2 measurements.
Fasting plasma glucose | Baseline and week 9
  Fasting plasma glucose will be measured from a fingerstick blood sample in the morning after an overnight fast using the Cholestech LDX System® (Hayward, CA).
Total Cholesterol | Baseline and week 9
  Total cholesterol will be quantified from a fingerstick blood sample in the morning after an overnight fast using the Cholestech LDX System® (Hayward, CA).
LDL Cholesterol | Baseline and week 9
  LDL cholesterol will be computed using the Friedewald equation from the lipid profile measured from a fingerstick blood sample in the morning after an overnight fast using the Cholestech LDX System® (Hayward, CA).
HDL Cholesterol | Baseline and week 9
  HDL cholesterol will be quantified from a fingerstick blood sample in the morning after an overnight fast using the Cholestech LDX System® (Hayward, CA).
Triglycerides | Baseline and week 9
  Triglycerides will be quantified from a fingerstick blood sample in the morning after an overnight fast using the Cholestech LDX System® (Hayward, CA).
Non-HDL Cholesterol | Baseline and week 9
  Non-HDL cholesterol will be computed by difference based on the lipid profile determined from a fasted fingerstick blood sample using the Cholestech LDX System® (Hayward, CA).
Resting heart rate | Baseline and week 9
  Resting heart rate will be measured in duplicate in the morning after 10 minutes of seated rest using Omron HEM-907XL Professional Digital Blood Pressure Monitors (Omron Healthcare, Kyoto, Japan).
Cardiorespiratory fitness based on post-exercise recovery heart rate | Baseline and week 9
  Cardiorespiratory fitness will be estimated based on heart rate recovery following a 3-minute step test performed with an 8-inch step and a metronome set to 96 beats/minute. Participants will be instructed to maintain the pace set by the beat of the metronome for 3 consecutive minutes and to be seated immediately at the completion of the 3-minute test. The subject's right radial pulse rate will be measured for 30 seconds, beginning 30 seconds after the completion of the test. Cardiorespiratory fitness level will be computed based on sex- and age-specific heart rate criteria.
Dietary patterns | Baseline and week 9
  Dietary patterns will be assessed using the nutrition questions from the CDC Behavioral Risk Factor Surveillance System (BRFSS).
Physical activity patterns | Baseline and week 9
  Physical activity patterns will be assessed using the exercise questions from the CDC Behavioral Risk Factor Surveillance System (BRFSS).
Perceived barriers to exercise participation | Baseline and week 9
  Perceived barriers to exercise participation will be assessed using the "Exercise Barriers" questionnaire, which the subject will complete on his/her own.
Perceived benefits of exercise | Baseline and week 9
  Perceived benefits of exercise will be assessed using the "Exercise Benefits" questionnaire, which the subject will complete on his/her own.
Participant evaluation of the wellness program | Weeks 12 - 14
  Participants will be asked to provide feedback about the wellness program through a 10-question, anonymous, online survey administered using the web-based Survey Monkey tool.

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Racette, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Result] Butler CE, Clark BR, Burlis TL, Castillo JC, Racette SB. Physical Activity for Campus Employees: A University Worksite Wellness Program. J Phys Act Health. 2015 Apr;12(4):470-6. doi: 10.1123/jpah.2013-0185. Epub 2014 Jun 4. PMID 24905703